CLINICAL TRIAL: NCT02672072
Title: Simulation-based Education for Managing Stress in ICU Nurses
Acronym: SISTRESSREA
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-04; RCAPHM15_0036 (Other: APHM)
Record Dates: First submitted 2016-01-22; First posted 2016-02-03 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-03

CONDITIONS: Professional Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control group: 5-day specific training with dedicated scenario done by an ICU expert simulation team after the period of the study
  Interventions: Other: questionnaire to define the presence of job strain at 6 months; Other: questionnaire to define the presence of job strain at 12 months
- Simulation group: 5-day specific training with dedicated scenario done by an ICU expert simulation team
  Interventions: Other: Simulation during the study (5-day specific training with dedicated scenario done by an ICU expert simulation team); Other: questionnaire to define the presence of job strain at 6 months; Other: questionnaire to define the presence of job strain at 12 months

INTERVENTIONS:
Other: Simulation during the study (5-day specific training with dedicated scenario done by an ICU expert simulation team)
  Groups: Simulation group
Other: questionnaire to define the presence of job strain at 6 months
Other: questionnaire to define the presence of job strain at 12 months

SUMMARY:
I. Main outcome Decrease of the stress evaluated 6 months after training. Stress is defined as the presence of job strain as defined by Karasek.

II. Main secondary outcomes

* ICU nurses stress at one year
* Burnout
* Intent-to-leave the ICU
* Quality of life

III. Design

Prospective, randomized, open study comparing 2 groups of ICU nurses:

Simulation group and Control group

Nurses from 9 different adult ICUs will be included. Stratification by ICU will be done (to take into account differences between the ICUs regarding organization, activity, patients…).

This study is observational because nurses can participate to this training when they want. The fact that nurses are in control group delays their participation to this training but does not forbid them to particpate. The nurses from control group will participate to training at the end of study.

IV. Specific measures Control group: none

Simulation group: 5-day specific training with dedicated scenario done by an ICU expert simulation team

V. Study duration 48 months

VI. Ethical aspects - Reglementary concerns

* Study accepted by the Comité Consultatif sur le Traitement de l'Information en matière de Recherche dans le domaine de la Santé (CCTIRS) and by the Commission Nationale de l'Informatique et des Libertés (CNIL)
* Information to the participants prior inclusion

VII. Study population Job strain evaluated in a French study was 59% . The same rate was observed in a survey done in our institution (Assistance Publique Hôpitaux de Marseille). We therefore hypothesized that the intervention (simulation) should be able to reduce the job strain from 59% to 45% of the participants. With a power of 80% and a risk a of 5%, this study needs to include 185 patients per arm. To take into account few participants who will not complete the study, we aimed to include a total of 400 ICU nurses.

VIII Results An interim analysis will be performed after 200 inclusions

ELIGIBILITY:
Inclusion Criteria:

* ICU nurses from adult ICUs with a professional experience in the actual ICU of at least 6 months and no decision to leave the ICU at the time of enrollment

Non inclusion Criteria:

* Less than 6 months of professional activity in the actual ICU at the time of enrollment
* Intent-to-leave in the next 6-month period
* Previous experience of this simulation program
* Pregnant women

Exclusion Criteria :

* ICU nurses who leave their city during the study period
* Pregnant women who miss their job during at least 4 weeks during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU nurses from adult ICUs with a professional experience in the actual ICU of at least 6 months and no decision to leave the ICU at the time of enrollment
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Presence of job stain evaluated by the French version of the Karasek scale | 6 months
  Presence of job strain: psychological demand of work > 21 and decision latitude < 72

SECONDARY OUTCOMES:
Stress evaluated by the Karasek scale | enrollment and 1 year
  Karasek questionnaire
Psychosocial risks (Copenhagen Psychosocial Questionnaire) | enrollment, 6 months and one year
  French version of the COPSOQ (Copenhagen Psychosocial Questionnaire)
Burnout (Maslach Burnout Inventory) | enrollment, 6 months and one year
  French version of the Maslach Burnout Inventory
Intent-to-leave (Number of enrolled nurses who leave the actual ICU) | enrollment, 6 months and one year
  Number of enrolled nurses who leave the actual ICU
Quality of life (visual analogic scale) | enrollment, 6 months and one year
  visual analogic scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM
Locations (1):
- AP-HM, Marseille, France

REFERENCES:
- [Derived] El Khamali R, Mouaci A, Valera S, Cano-Chervel M, Pinglis C, Sanz C, Allal A, Attard V, Malardier J, Delfino M, D'Anna F, Rostini P, Aguilard S, Berthias K, Cresta B, Iride F, Reynaud V, Suard J, Syja W, Vankiersbilck C, Chevalier N, Inthavong K, Forel JM, Baumstarck K, Papazian L; SISTRESSREA Study Group. Effects of a Multimodal Program Including Simulation on Job Strain Among Nurses Working in Intensive Care Units: A Randomized Clinical Trial. JAMA. 2018 Nov 20;320(19):1988-1997. doi: 10.1001/jama.2018.14284. PMID 30357264